CLINICAL TRIAL: NCT07380061
Title: Feasibility and Preliminary Effectiveness of a Bidirectional Peer - Mentor Text Messaging Intervention to Promote Perinatal Mental Health: A Pilot Randomized Trial
Brief Title: Peer Mentor Texting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Amritha Subray Bhat, Associate Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00013616
Record Dates: First submitted 2026-01-06; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Perinatal Depression; Perinatal Anxiety; Parenting Stress
Keywords: perinatal mental health; text messaging; peer support

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): If assigned to Nurture (intervention arm), the participant was matched with a mentor from Nurture based on participants responses in their intake form which asked if there was anything in particular that they wanted support with and if there were characteristics that were important to them to share with their mentor. The mentor sent weekly messages based on a library of prompts. Prompts provided resources on child development, connections to local support agencies, and suggestions for parent-child bonding and parental wellness activities.
  Interventions: Behavioral: Peer mentor texting
- Control (Active Comparator): Participants receive automated interventional texts
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Peer mentor texting — If assigned to Nurture (intervention arm), the participant was matched with a mentor from Nurture based on participants responses in their intake form which asked if there was anything in particular that they wanted support with and if there were characteristics that were important to them to share with their mentor. The mentor sent weekly messages based on a library of prompts. Prompts provided resources on child development, connections to local support agencies, and suggestions for parent-child bonding and parental wellness activities.
  Arms: Intervention
Behavioral: Control — If assigned to the control arm, the participant received automated informational texts throughout the period of participation. Participants could not respond to these texts. Information content that is publicly available such as the Babycenter's pregnancy stage information the Washington State Department of Children, Youth, and Families (DCYF) information packets about infant development and milestones as well as various ways to encourage learning and healthy development was used.
  Arms: Control

SUMMARY:
This study tested whether a peer mentor text message program (called the Nurture program) could help support mental health during pregnancy and after birth. In the study, 127 pregnant people in Washington state were randomly placed to in one of two groups: Nurture group - could text with a trained peer mentor and Control group got automated informational text messages. Researchers looked at how much participants used the program and whether it affected symptoms of depression, anxiety and stress related to parenting. Most people in the Nurture group actively used the program. Nearly all responded to their mentor and there was an average of 32 back and forth text conversations. Mentors usually started more conversations than participants did. People using Nurture had lower anxiety six weeks after giving birth compared to the control group. However there were no statistically significant differences between the two groups for depression or parenting stress. The findings suggest that having two way text conversations with peer mentors is well received and may help reduce anxiety soon after birth. More research with larger groups is needed to understand the full benefits and how to make the program widely available.

ELIGIBILITY:
Inclusion Criteria:

* Women and other birthing individuals receiving prenatal care within Washington.

Exclusion Criteria:

* Severe mental illness such as bipolar disorder and schizophrenia and severe substance use disorder based on self report.
* Severe depression symptomology operationalized as PHQ-9 score 20 or higher.
* Severe suicidality (a response of "Nearly every day" to question 9, "Over the last 2 weeks, how often have you been bothered by any of the following problems?: Thoughts that you would be better off dead or of hurting yourself in some way." on the PHQ-9 questionnaire.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-05-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline in depressive symptoms over time as measured by the PHQ-9 | Baseline, 6 weeks, 3 months, 6 months and 9 months postpartum.
  Depressive symptoms in pregnancy and postpartum measured using the Patient Health Questionnaire -9 (PHQ-9). Score range 0 to 27, with higher scores meaning worse depression.
Change from baseline in anxiety symptoms over time, as measured by GAD-7. | Baseline, 6 weeks, 3 months, 6 months and 9 months postpartum.
  Anxiety during pregnancy and postpartum, measured using the Generalized Anxiety disorder Scale (GAD-7). Score range from 0 to 27 with higher scores meaning worse anxiety
Change from baseline to 9 months in Parenting Stress as measured by the Parenting Stress Scale | 6 weeks and 9 months postpartum.
  Parenting Stress measured using the Parenting Stress Scale. An 18 - item self report scale - items represent positive (e.g. emotional benefits, personal development) and negative (demands on resources, restrictions) themes of parenthood. Overall possible scores on the scale range from 18 - 90. The higher the score , the higher the measured level of Parental stress
Feasibility of enrolment as measured by number of participants enrolled | Baseline
  Ability to enroll into the study
Intervention engagement as measured by number of messages exchanged | Baseline, 9 months postpartum
  Engagement measured by number of messages exchanged

SECONDARY OUTCOMES:
Change from baseline in General Wellbeing over time as measured by the General Wellbeing Schedule | Baseline, 6 weeks, 3 months, 6 months and 9 months postpartum.
  Measure of wellbeing, score range 0 - 110, higher scores indicating higher wellbeing.
Change in Maternal self efficacy from baseline over time as measures by the Self Efficacy in a Nurturing Role questionnaire. | Baseline, 6 weeks and 9 months postpartum.
  Parenting self efficacy measured during pregnancy and postpartum, using the Self Efficacy in a Nurturing Role questionnaire.16 items, score range 16 - 112, higher scores represent higher self efficacy.
Change in wellbeing from baseline to 9 months as measured by the Flourishing scale | Baseline and 9 months postpartum.
  Measure of wellbeing. Score range is 8 to 56, with higher scores representing a person with many psychological resources and strengths.
Social support | Baseline, 3 months and 9 months postpartum.
  Social support measured using Multidimensional scale of perceived social support (MSPSS). The MSPSS a 12-item self-report questionnaire that measures perceived support from family, friends, and significant others.
  Score Range 12 to 84, low scores indicating low support and high scores indicating high support.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No